CLINICAL TRIAL: NCT06462053
Title: A Prospective, Randomized, Phase II Trial of Short-course Radiotherapy Combined With CAPOX and PD-1 Antibody Versus Long-course Chemoradiotherapy Combined With CAPOX for Early Low-lying Rectal Cancer
Brief Title: Short-course Radiotherapy Combined With CAPOX and PD-1 Antibody Versus Long-course Chemoradiotherapy Combined With CAPOX for Early Low-lying Rectal Cancer
Acronym: TORCH-E2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2023-377-3496
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Early Low Rectal Cancer
MeSH Terms: interventions — toripalimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-course Radiotherapy plus immunochemotherapy group (Experimental): The patients will receive short-course radiotherapy (25Gy/5Fx, SCRT), followed by 4 cycles of CAPOX and PD-1 antibody, finally receive the TEM or TME surgery or adopt WW option.
  Interventions: Radiation: Short-course radiotherapy; Drug: PD-1 antibody (Toripalimab); Drug: Oxaliplatin; Drug: Capecitabine
- Long-course Radiotherapy plus chemotherapy group (Experimental): The patients will receive long-course radiotherapy (50Gy/25Fx,LCRT, concurrent capecitabine), followed by 2 cycles of CAPOX, finally receive the TEM or TME surgery or adopt WW option.
  Interventions: Radiation: Long-course radiotherapy; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Radiation: Short-course radiotherapy — Short-course radiotherapy: 25Gy/5Fx
  Other Names: SCRT
  Arms: Short-course Radiotherapy plus immunochemotherapy group
Drug: PD-1 antibody (Toripalimab) — Toripalimab 240mg d1 q3w
  Other Names: Toripalimab
  Arms: Short-course Radiotherapy plus immunochemotherapy group
Radiation: Long-course radiotherapy — Long-course radiation: 50Gy/25Fx
  Other Names: LCRT
  Arms: Long-course Radiotherapy plus chemotherapy group
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w
Drug: Capecitabine — Xeloda
  Other Names: Xeloda

SUMMARY:
TORCH-E2 is a prospective, multicentre, randomized phase II trial. 134 low-lying early (T1-3b/N0-1M0, distance from anal verge ≤5cm) patients will be recruited and assigned to Group 1 and Group 2 (1:1). Group 1 receives SCRT (25Gy/5Fx) followed by 4 cycles of capecitabine plus oxaliplatin (CAPOX) chemotherapy and PD-1 antibody. Group 2 receives LCRT (50Gy/25Fx) followed by 2 cycles of CAPOX. A WW option can be applied to patients achieving cCR while surgery will be recommended for those who fail to achieve cCR. The primary endpoint is complete response (CR, pathological complete response [pCR] plus cCR) rate. The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, anal preservation rate, 3-year DFS rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years old, female and male
2. pathological confirmed adenocarcinoma
3. clinical stage T1-3bN0-1, tumor maximum diameter less than 4cm
4. the distance from anal verge less than 5 cm
5. without distance metastases
6. KPS >=70
7. with good compliance
8. microsatellite repair status is MSS/pMMR
9. without previous anti-cancer therapy or immunotherapy
10. signed the inform consent

Exclusion Criteria:

1. pregnancy or breast-feeding women
2. pathological confirmed signet ring cell carcinoma
3. clinical stage T1N0 and can be resected locally
4. history of other malignancies within 5 years
5. serious medical illness, such as severe mental disorders, cardiac disease, uncontrolled infection, etc.
6. immunodeficiency disease or long-term using of immunosuppressive agents
7. baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
8. DPD deficiency
9. allergic to any component of the therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | 1 month after the surgery or the decision of W&W
  Rate of complete response (CR), including the rate of pathologic complete response (pCR) after surgery and the rate of cCR with W&W strategy.

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From date of randomization until 3 months after the completion neoadjuvant therapy
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
Organ preservation rate | from date of receiving neoadjuvant therapy, assessed up to 3 years
  Organ preservation rate
3 year disease free survival rate | From date of initiation of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Rate of 3 year disease free survival
3 year local recurrence free survival rate | From date of initiation of treatment until the date of first documented pelvic failure, assessed up to 36 months.
  Rate of 3 year local recurrence free survival
3 year overall survival rate | From date of initiation of treatment until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
3 year Quality of Life | From date of initiation of treatment until the date of death from any cause, assessed up to 3 years
  Quality of life will be evaluated using EORTC QLQ-C30, EORTC QLQ-CR29, LARS score and Wexner score.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, M.D, PH.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China